CLINICAL TRIAL: NCT05964647
Title: Effect of Ketanserin, Olanzapine, and Lorazepam After LSD Administration on the Acute Response to LSD in Healthy Subjects
Acronym: LBL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BASEC ID 2023-01075
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: LSD; Serotonin; Psychedelics
MeSH Terms: interventions — Lysergic Acid Diethylamide; Ketanserin; Olanzapine; Lorazepam

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LSD + ketanserin (Active Comparator)
  Interventions: Drug: LSD (150 µg) + ketanserin (40 mg)
- LSD+ olanzapine (Active Comparator)
  Interventions: Drug: LSD (150 µg) + olanzapine (10 mg)
- LSD+ lorazepam (Active Comparator)
  Interventions: Drug: LSD (150 µg) + lorazepam (2 mg)
- LSD + placebo (Active Comparator)
  Interventions: Drug: LSD (150 µg) + placebo
- Placebo + placebo (Placebo Comparator)
  Interventions: Drug: Placebo + placebo

INTERVENTIONS:
Drug: LSD (150 µg) + ketanserin (40 mg) — Drug: LSD (150 µg) per os, single dose
  Other: Ketanserin (40 mg) per os, single dose
  Arms: LSD + ketanserin
Drug: LSD (150 µg) + olanzapine (10 mg) — Drug: LSD (150 µg) per os, single dose
  Other: Olanzapine (10 mg) per os, single dose
  Arms: LSD+ olanzapine
Drug: LSD (150 µg) + lorazepam (2 mg) — Drug: LSD (150 µg) per os, single dose
  Other: Lorazepam (2 mg) per os, single dose
  Arms: LSD+ lorazepam
Drug: LSD (150 µg) + placebo — Drug: LSD (150 µg) per os, single dose
  Other: Placebo (Capsules containing mannitol looking identical to the other drugs)
  Arms: LSD + placebo
Drug: Placebo + placebo — Drug: Placebo (Capsules containing mannitol looking identical to the other drugs)
  Other: Placebo (Capsules containing mannitol looking identical to the other drugs)
  Arms: Placebo + placebo

SUMMARY:
The main objective of this study is to determine whether administration of ketanserin (40 mg), olanzapine (10 mg), and lorazepam (2 mg) after administration of LSD (150 µg) attenuates and shortens the subjective LSD response (any drug effect) compared to administration of LSD (150 µg) alone

DETAILED DESCRIPTION:
LSD is investigated as treatment for various psychiatric (e.g., depression and anxiety) but also somatic disorders (e.g., cluster headache). In Switzerland, compassionate use of psychedelics including LSD is possible based on single authorizations of the federal office of public health in treatment-resistant patients. Additionally, current social and political changes demonstrate a shift of how psychedelics are seen and how they might be used in therapy in the future.

Despite the good safety profile of LSD, a broader use might increase the number of adverse psychological reactions to LSD. For such occasions, health professionals should have a tool to not only psychologically but also pharmacologically interfere and end states of acute psychedelic-induced distress. In clinical practice, the gamma-butyric acid (GABA) agonistic acting benzodiazepine lorazepam or the atypical neuroleptic olanzapine with affinity to the 5-HT2A, 5-HT2C and dopamine D1-4 receptors are primarily used for the treatment of drug-induced psychotic symptoms. However, the ability of these drugs to block these effects after LSD intake remains to be investigated.

The primary goal of the present study is therefore to investigate whether ketanserin, olanzapine and lorazepam administration after LSD administration might attenuate and shorten the LSD response compared to administration of LSD alone. Additionally, the present study examines changes in quality of the LSD experience after administration of ketanserin, olanzapine or lorazepam and effects on sensorimotor gating and sleep. The study provides insight into the receptor mechanisms involved in alterations of consciousness and specifically the relevance of ongoing 5-HT2A receptor stimulation in the mediation of the psychedelic response to LSD and psychotic symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids and foods from the evenings prior to the study sessions to the end of the study days, limit coffee drinking ≤ 3 cups per day for 7 days prior to study day
7. Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration
8. Willing to use effective contraceptive measures throughout study participation (according to Clinical Trial Facilitation Group (CTFG): Recommendations related to contraception and pregnancy testing in clinical trials)
9. Women of childbearing potential must have a negative pregnancy test at the beginning of the study. Pregnancy tests are repeated before each study session.
10. Body mass index between 18 - 29 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder including psychotic disorder, mania / hypomania, borderline personality disorders.
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Known hypersensitivity to LSD, ketanserin, olanzapine or lorazepam
5. Hypertension (>140/90 mmHg) or hypotension (SBP < 85 mmHg)
6. Hallucinogenic substance use (not including cannabis) more than 10 times or any time within the previous two months
7. Pregnancy or current breastfeeding
8. Participation in another clinical trial (currently or within the last 30 days)
9. Use of medication that may interfere with the effects of the study medication
10. Current substance use disorder (within the last 2 months)
11. Tobacco smoking (>1 cigarette/day)
12. Consumption of alcoholic beverages (>15 drinks/week)
13. Not exhibiting consistent startle responding on the screening day (i.e., over 75% discernible responses to six 108 dB 40 ms startle pulses), as this would preclude the ability to measure fear potentiated startle.
14. Use of strong CYP2D6 inhibitor
15. Use of strong CYP1A2 inhibitor or inducer

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Duration of subjective response | 18 months
  Visual Analog Scales (VAS) will be repeatedly used to assess subjective alterations in consciousness over time. VAS will be presented as 100 mm long horizontal lines marked with: "not at all" on the left and any drug effect", "good drug effect", "bad drug effect", "stimulated", "tiredness", "fear", "nausea", "alteration of vision", "alteration of hearing", "sounds seem to influence what I see", "alteration of sense of time", "the boundaries between myself and my surroundings seem to blur", "I gain insights into contexts that were previously mysterious to me", "opposites dissolve", "talkative", "happy", and "trust". Additionally, "my perception is…" from "muted" to "clear", "I feel …" from "relaxed" to "tense", and "I feel my thoughts are …" from "sluggish" to "racing". Subjects will mark the scale with vertical lines.
Extent of subjective response | 18 months
  Area under the curve (AUEC), Emax, of the VAS-Item "any drug effect"

SECONDARY OUTCOMES:
Alterations of consciousness | 18 months
  Altered States of Consciousness 5 Dimensions of Altered States of Consciousness (5D-ASC) assesses mood, anxiety, derealization, depersonalization, changes in perception, auditory alterations, and reduced vigilance. The questionnaire is consisting of 94 items to be rated on a visual analog scale (horizontal line, 100 mm, marked with "not at all" on the left and "extremely" on the right), with higher values indicating stronger effects. Subjects will mark the scale with vertical lines.
Mystical-type effects | 18 months
  Mystical-type experience questionnaire (MEQ) assesses with 30 items (embedded into the SCQ) the mystical experiences on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely").
Subjective effects I | 18 months
  Visual Analog Scales (VAS) will be repeatedly used to assess subjective alterations in consciousness over time. VAS will be presented as 100 mm long horizontal lines marked with: "not at all" on the left and any drug effect", "good drug effect", "bad drug effect", "stimulated", "tiredness", "fear", "nausea", "alteration of vision", "alteration of hearing", "sounds seem to influence what I see", "alteration of sense of time", "the boundaries between myself and my surroundings seem to blur", "I gain insights into contexts that were previously mysterious to me", "opposites dissolve", "talkative", "happy", and "trust". Additionally, "my perception is…" from "muted" to "clear", "I feel …" from "relaxed" to "tense", and "I feel my thoughts are …" from "sluggish" to "racing". Subjects will mark the scale with vertical lines.
Subjective effects II | 18 months
  Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely".
Subjective effects III | 24 hours
  The Addiction Research Center Inventory (ARCI) is a true-false questionnaire with five empirically derived scales. The scale is administered once before, after 3 h, 10 h, and 24 h after LSD administration.
Psychotomimetic effects I | 18 months
  The aberrant salience inventory (ASI) is a 29-item questionnaire rated as "yes" or "no" measuring trait aberrant salience, which has been hypothesized to be important for psychosis and psychotic disorders. The questionnaire will be administered once at the end of the session and subjects will be instructed to retrospectively rate peak alterations during the study session.
Psychotomimetic effects II | 18 months
  The psychotomimetic states inventory (PSI) consists of 48 items measuring "psychosis-like" experiences and is one of the most widely used measure of drug-induces psychotic-like effects. Items will be scored on a 4-point scale (0 = never to 3 = strongly). The questionnaire will be administered once at the end of the session and subjects will be instructed to retrospectively rate peak alterations during the study session.
Effects of LSD on mindfulness and decentering I | 36 hours
  The 39-item Five Facet Mindfulness Questionnaire (FFMQ) measures five facets of a general tendency to be mindful in daily life. The FFMQ will be completed by the participants at screening, the beginning of each study session (to assess respective baseline) and will be handed in to the participants at the end of the respective study visit and participants will be asked to complete the FFMQ at home 36 h after the study drug has been administered.
Effects of LSD on mindfulness and decentering II | 36 hours
  The 20-item Experience Questionnaire (EQ) measures decentering and ruminating. Decentering is defined as looking at one's own feelings from a distance, in an observing and objective way. The EQ will be completed by the participants at screening, at the beginning of each study session (to assess respective baseline) and will be handed in to the participants at the end of the respective study visit, and participants will be asked to complete the EQ at home 36 h after the study drug has been administered
Challenging experiences | 18 months
  The Challenging Experiences Questionnaire (CEQ) was developed to characterize challenging experiences with psilocybin. The 26-item questionnaire is rated on a 6-point Likert scale ranging from 0 (none, not at all) to 5 (extreme, more than ever before in my life). The CEQ includes seven factors: "Fear"; "Grief"; "Physical Distress"; "Insanity"; "Isolation"; "Death"; "Paranoia", and a total score (Total) is calculated over all items. 9. The validated German version of the CEQ 153 will be administered once at the end of the session and subjects will be instructed to retrospectively rate their experiences during peak alterations during the study session.
Effects on prepulse inhibition and sensorimotor gating | 18 months
  Prepulse inhibition (PPI) of the acoustic startle response is an operational measure of sensorimotor gating that can be measured in animals and humans and serves as a preclinical model for schizophrenia. LSD and other serotonergic 5-HT2A agonists disrupt PPI in animals and in humans and PPI is also disrupted in schizophrenic patients. We will measure effects of LSD on sensorimotor gating function.
Blood pressure | 18 months
  Blood pressure, assessed 21 times during each study session via systolic and diastolic blood pressure.
Heart rate | 18 months
  Heart rate, assessed 21 times during each study session via heart rate, Emax.
Body temperature | 18 months
  Body temperature assessed 20 times during each study session via tympanic body temperature.
Pupil size | 18 months
  Pupil size, assessed 8 times during each study session via pupilometer.
LSD concentrations in the blood | 18 months
  LSD and metabolites concentrations measured in the blood plasma, assessed 17 times during each study session via blood samples.
Ketanserin concentrations in the blood | 18 months
  Ketanserin concentrations measured in the blood plasma, assessed 17 times during each study session via blood samples.
Olanzapine concentrations in the blood | 18 months
  Olanzapine concentrations measured in the blood plasma, assessed 17 times during each study session via blood samples.
Lorazepam concentrations in the blood | 18 months
  Lorazepam concentrations measured in the blood plasma, assessed 17 times during each study session via blood samples.
Effects of LSD on sleep phases | 11 hours
  The Dreem® headband will record electroencephalographic (EEG; five dry electrodes yielding seven derivations), acceleration (3D accelerometer), and heart rate (red-infrared pulse oximeter) activity. We will further calculate sleep variables of %REM (REM sleep duration divided by total sleep duration), REM Latency (duration of non-REM sleep before the first REM phase), and REM Efficiency (REM sleep duration divided by the total REM episode duration) for each night. We will start the measurement 11 h after LSD administration until the end of the study day.
Persisting effects | 18 months
  The 143-item Johns Hopkins University Persisting Effects Questionnaire (PEQ) seeks information about changes in attitude, mood, behavior, and spiritual experience items are rated on a six-point scale. The PEQ will be administered at the EOS visit.
Adverse effects | 18 months
  The adapted list of complaints (LC) consists of 50 items offering a global score measuring physical and general discomfort. The LC list is administered before, 12 h after LSD administration with reference to all complaints arising since the LSD administration, and at the end of the session with reference to complaints throughout the night. Subjects will additionally be asked to report any adverse events during the sessions or/and between study sessions as assessed at the beginning of the next session and at the EOS visit.
Emotional effects | 18 months
  Multifaceted Empathy Test (MET), effects on empathy in computer tests, assessed one time during each study session.
Sleepiness | 18 months
  The Karolinska Sleepiness Scale (KSS) measures the subjective level of sleepiness 161. The scale shows a 10-point scale from "1 - extremely alert" to "10 - extremely sleepy - cannot stay awake". The KSS will be assessed at the beginning and repeatedly in the evening and next morning of the study session
Effect moderation through personality traits I | 18 months
  Assessed one time during the screening via the NEO-Five-Factor-Inventory (NEO-FFI). The NEO-FFI assesses 5 personality traits (openness to experience, conscientiousness, extraversion, agreeableness and neuroticism) consisting of of 60 items. Each item is evaluated on a scale from -- "strong disagreement" to ++ "strong agreement".
Effect moderation through personality traits II | 18 months
  Assessed one time during the screening via Freiburger Personality Inventory (FPI). The FPI-R version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Effect moderation through personality traits III | 18 months
  Assessed one time during the screening via Saarbrücker Personality Questionnaire (SPF). The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
Effect moderation through personality traits IV | 18 months
  Assessed one time during the screening via HEXACO personality inventory (Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness, and Openness). The HEXACO consists of 100 items. Each item is evaluated on a scale from 1 "strong disagreement" to 5 "strong agreement".
Effect moderation through personality traits V | 18 months
  Assessed one time during the screening via Defense Style Questionnaire (DSQ-40). The DSQ-40 can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No